CLINICAL TRIAL: NCT06562218
Title: The Effectiveness of Cross-training on an Immobilised Forearm Due to Fracture
Brief Title: The Effectiveness of Cross-training on an Immobilised Forearm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dilara Ekici Zincirci (Other)
Responsible Party: Sponsor-Investigator, Dilara Ekici Zincirci, Medical Doctor, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Organization: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CTO-CE1
Record Dates: First submitted 2024-08-16; First posted 2024-08-20 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2024-11

CONDITIONS: Forearm Fracture
Keywords: fracture; immobilisation; cross-education; muscle strength
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Intervention Model Description: prospective randomized controlled double-blind clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not know which group they have been assigned to, and the researchers evaluating the results will not know which group participants have been assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- cross training group (Experimental): Group whose healthy arm (unbroken side) is strengthened
  Interventions: Procedure: isokinetic strengthening exercise
- control group (Experimental): group given conventional exercise to the fractured arm
  Interventions: Procedure: conventional exercise programm

INTERVENTIONS:
Procedure: isokinetic strengthening exercise — Participants' isokinetic strength measurements will be assessed using the Cybex II Humac Norm isokinetic dynamometer. A strengthening programme will be performed for a total of 12 sessions, 3 days a week for 4 weeks, at 20 degrees of flexion, 20 degrees of extension, 60-90 and 180 degrees/s speed.
  At the beginning and end of the 12th session, isokinetic and isometric muscle performance tests will be performed on the healthy wrist, and isometric wrist flexor and extensor strength measurements will be performed in neutral position 1 week after removal of the cast on the fractured wrist.
  Arms: cross training group
Procedure: conventional exercise programm — The immobilised limb was given finger grip exercises.
  Arms: control group

SUMMARY:
The cross-training phenomenon is the increase in muscle strength in the contralateral limb when one limb is exercised. Limited studies have shown that it prevents immobilisation-induced muscle weakness in healthy volunteers. The aim of this study was to evaluate the effect of strengthening the contralateral extremity on muscle strength and range of motion in the immobilised extremity in patients who had undergone immobilisation for forearm fractures.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic unilateral forearm fracture (treated surgically or conservatively and immobilised in a cast)

Exclusion Criteria:

* Previous upper limb surgery/joint disease - deformity affecting hand-wrist function
* Any neurological condition affecting the upper extremity (stroke, Parkinson's disease; multiple sclerosis, reflex sympathetic dystrophy, peripheral nerve injury)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-08-26 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Wrist isometric flexion muscle strength | 1 year
  The isometric flexion strength of the fractured wrist will be measured using an isokinetic dynamometer at the first week after immobilisation has ceased.
Wrist isometric extansion muscle strength | 1 year
  The isometric extansion strength of the fractured wrist will be measured using an isokinetic dynamometer at the first week after immobilisation has ceased.

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Dr. Cemil Taşçıoğlu City Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No